CLINICAL TRIAL: NCT01381601
Title: Incidence, Prevalence, and Symptom Burden Associated With Advanced Renal Cell Carcinoma in Commercially Insured Population (Pharmetrics)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114866
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Carcinoma, Renal Cell
Keywords: retrospective database analysis; economic burden
MeSH Terms: conditions — Carcinoma, Renal Cell; Financial Stress | interventions — Sunitinib; Sorafenib; Bevacizumab; pazopanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe adverse event claims in subjects with metastatic RCC: Presence or absence of common severe treatment related adverse events (based on existence of claims) in patients with metastatic RCC. Common severe adverse event defined as Grade 3 or higher with >=5% frequency of occurence as reported in product label.
  Interventions: Drug: Targeted agents indicated in management of advanced/metastatic RCC (sunitinib, sorafenib, bevacizumab, and pazopanib)

INTERVENTIONS:
Drug: Targeted agents indicated in management of advanced/metastatic RCC (sunitinib, sorafenib, bevacizumab, and pazopanib) — Metastatic RCC patients on either sunitinib or sorafenib or bevacizumab or pazopanib (identified based on claims) will be evaluated for presence or absence of common severe adverse events. These common severe adverse events will be identified from agent's product labels.
  Other Names: VOTRIENT™ (pazopanib); SUTENT® (sunitinib malate); AVASTIN® (bevacizumab); NEXAVAR® (sorafenib)

SUMMARY:
Information on the prevalence of advanced/metastatic renal cell carcinoma and its symptom burden is limited in commercially insured adult patients. Additionally, limited information exists on economic burden of adverse events associated with treatments for advanced/metastatic renal cell carcinoma. An objective of the current study is to estimate the incidence, prevalence, and symptom burden associated with advanced/metastatic RCC in a US "real-world" setting. Another objective is to quantify the economic burden of severe adverse events with agents used in management of first line advanced/metastatic RCC (sunitinib, sorafenib, bevacizumab, and pazopanib). This study will employ a retrospective cohort design. Analyses of health insurance claims data from a large commercially insured population will be employed in the current study. Study subjects will consist of all persons, aged ≥18 years, with evidence of advanced RCC between January 1, 2000 and December 31, 2009; these persons will be identified based in part on case-ascertainment algorithms. Analyses will be directed at estimating annual rates of incidence and prevalence of advanced/metastatic RCC, as well as symptom burden and costs of common severe adverse events associated with treatments used in management of advanced/metastatic RCC (sunitinib, sorafenib, bevacizumab, and pazopanib).

ELIGIBILITY:
Inclusion Criteria:

* two or more medical encounters with a diagnosis of kidney cancer (ICD-9-CM 189.0) or malignant neoplasm of the renal pelvis (189.1), and
* two or more medical encounters with a diagnosis of distant secondary malignant neoplasm (ICD-9-CM 197.XX-199.0, excluding 198.0 [kidney metastasis]) on different days <120 days apart (the date of the earliest such encounter will be designated the "index date").

Exclusion Criteria:

* evidence of receipt of chemotherapeutic agents indicated or used in the treatment of advanced TCC, or
* evidence of cystoscopy, biopsy of the bladder, or radical cystectomy
* evidence of any other primary cancer

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study subjects will be selected from a source population consisting of all persons in the PharMetrics database with one or more days of eligibility for comprehensive health benefits between January 1, 2000 and December 31, 2009.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
New and existing claims of metastatic renal cell carcinoma across multiple years | 2000 - 2009 (up to 10 years)
  Identifying new and existing claims (based on claims based case-ascertainment algorithm) of metastatic renal cell carcinoma across multiple years
Cost associated with management of common severe adverse events related to 1st line treatments used in metastatic renal cell carcinoma | 2000 - 2009 (up to 10 years)
  Quantifying economic burden associated with management of common severe adverse events (defined as grade 3 and above adverse events occurring >= 5% as per product label) related to agents used in 1st line metastatic RCC (sunitinib, sorafenib, bevacizumab, and pazopanib). Adverse events will be identified based on product labels.

SECONDARY OUTCOMES:
Quantify symptom burden associated with metastatic renal cell carcinoma | 2000 - 2009 (up to 10 years)
  Quantifying symptom burden based on identification of claims associated with the respective symptoms. Disease related symptoms will be identified based on published literature.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline